CLINICAL TRIAL: NCT02084927
Title: Hyperbaric Oxygen Therapy Can Improve Neurological State Post Meningioma Removal Surgery -Randomized Prospective Trial
Brief Title: Hyperbaric Oxygen Therapy Can Improve Neurological State Post Meningioma Removal Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Shai Efrati, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 37/14
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Intracranial Meningioma; Neurologic Deficits
MeSH Terms: conditions — Meningioma; Neurologic Manifestations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HBOT (Experimental): Group will be treated with HBOT for 60 treatments in 3 months.
  Interventions: Biological: HBOT
- Control/Crossover (Other): Control for 3 months without treatment, and then HBOT for 60 treatments in 3 months.
  Interventions: Biological: HBOT

INTERVENTIONS:
Biological: HBOT — HBOT of 2 ATA for 90 minutes, for 60 treatments

SUMMARY:
The aim of the current study is to evaluate, in a prospective cross-over, randomized study, the effect of hyperbaric oxygen therapy (HBOT) on patients with chronic neurological deficits and cognitive impairment after anterior skull base meningioma tumor removal.

ELIGIBILITY:
Inclusion Criteria:

* Post intracranial meningioma removal surgery 3-12 months prior to the inclusion in the study.
* All patients have to have persistent cognitive or neurological complaints regarding without noticeable improvement during the last month prior to their enrolment.
* Age 18 years or older.

Exclusion Criteria:

* Dynamic neurologic/cognitive improvement or worsening during the past month;

  * Evidence of dynamic cognitive/neurological improvement in the last month.
  * Previous brain radiotherapy and/or radiosurgery.
  * Steroids dependence
  * Seizures 1 month previous to inclusion
  * Had been treated with HBOT for any other reason 1 month prior to inclusion;
  * Have any other indication for HBOT;
  * Chest pathology incompatible with pressure changes;
  * Inner ear disease;
  * Patients suffering from claustrophobia;
  * Inability to sign written informed consent;
  * Smoking patients will not be allowed to smoke during the study and if they would not comply with this demand they will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive functions | 6 months
  Cognitive function will be assessed using the one-hour Mindstreams Computerized Cognitive Test Battery at baseline, 3 months and 6 months to intervention.

SECONDARY OUTCOMES:
Quality of Life | 6 months
  Quality of live will be evaluated by the EQ-5D questionnaire at baseline , 3 months and 6 months to intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Study Chair — Assaf-Harofeh Medical Center
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel